CLINICAL TRIAL: NCT04147013
Title: Effect of Celecoxib on Postoperative Narcotic Use and Disease Severity in Patients with Aspirin-exacerbated Respiratory Disease and Chronic Rhinosinusitis: a Randomised Controlled Trial
Brief Title: Effect of Celecoxib on Postoperative Analgesia and Disease Severity in AERD Patients with CRS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114809
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Chronic Rhinosinusitis with Nasal Polyps; Aspirin-exacerbated Respiratory Disease
Keywords: Analgesia; Analgesic opioids; Nasal Polyposis; Treatment
MeSH Terms: conditions — Agnosia; Nasal Polyps | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: A prospective, double-blinded, randomized controlled study.
Who Masked: Participant, Investigator
Masking Description: The control group will use a placebo pill, instead of an active drug. The randomization process will be held by the Site's Pharmacy. Hence, the investigators will only have access to a list of randomized numbers, associated with the available drug/placebo pills, to implement during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib Group (Experimental): Patients will receive the interventional drug for 7 days post endoscopic sinus surgery. These patients will also receive a prescription for tramadol (50 mg PO Q6H PRN x 10 tablets), to be used as needed for breakthrough pain. Patients will also be permitted to take acetaminophen for breakthrough pain as needed and will be encouraged to use acetaminophen prior to narcotic usage. Finally, they will be prescribed a nasal saline rinse, which is to be started on postoperative day one.
  Interventions: Drug: Celecoxib
- Control Group (Placebo Comparator): Patients will receive the placebo for 7 days post endoscopic sinus surgery. These patients will also receive a prescription for tramadol (50 mg PO Q6H PRN x 10 tablets), to be used as needed for breakthrough pain. Patients will also be permitted to take acetaminophen for breakthrough pain as needed and will be encouraged to use acetaminophen prior to narcotic usage. Finally, they will be prescribed a nasal saline rinse, which is to be started on postoperative day one.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Patients will receive celecoxib 200 mg PO BID for 7 days post endoscopic sinus surgery, starting on the evening of the day of surgery.
  Other Names: Celebrex
  Arms: Celecoxib Group
Drug: Placebo — Patients will receive placebo PO BID for 7 days post endoscopic sinus surgery, starting on the evening of the day of surgery.
  Arms: Control Group

SUMMARY:
This is a proposed randomized prospective study to evaluate both the anti-inflammatory and analgesic effects of a COX-2 inhibitor, celecoxib, in patients with aspirin-exacerbated respiratory disease and Chronic rhinosinusitis following endoscopic sinus surgery.

The investigators hypothesize that supplementation with celecoxib can potentially improve surgical outcomes and reduce the postoperative usage of opioid analgesics without an increased risk of bleeding or asthma exacerbation

DETAILED DESCRIPTION:
1. Background: Chronic rhinosinusitis (CRS) affects up to 5% of Canadians and is associated with significant morbidity. It is characterized by inflammation of the mucosa of the nose and paranasal sinuses of at least 12 consecutive weeks' duration. Patients suffering from CRS are bothered on a daily basis by nasal obstruction, nasal discharge, facial pain, and an impaired sense of smell among other symptoms. Although not typically a life-threatening condition, CRS can drastically reduce a patient's quality of life as well as their workplace productivity. In fact, this has been demonstrated in the literature, with one study estimating the annual productivity cost of refractory CRS at about $10,000 per patient.

   Fortunately, effective management strategies are available. Mild to moderate disease can often be managed safely with long term use of topical glucocorticoids and nasal saline lavage. For more severe CRS unresponsive to appropriate medical therapy, oral glucocorticoids can be effective in the short term, but surgical treatment can help achieve long-term control of symptoms when initial medical therapy has failed. This is typically done via endoscopic sinus surgery (ESS), and its goal is to re-establish physiological patterns of ventilation and mucociliary clearance in patients with CRS, as well as establish access for topical therapy delivery. ESS is considered the gold standard of management for CRS and has proven to be highly effective in reducing the burden of inflammatory tissue and minimizing patient morbidity.

   Although developed as a minimally invasive technique to avoid the morbidity of open sinus surgery, ESS still entails some degree of surgical trauma, postoperative pain, and inflammation. Intraoperative local anesthetic infiltration is routinely performed but is insufficient to control pain in the immediate postoperative period. Patients often require some form of systemic analgesia and this usually consists of some combination of acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen, and opioids. However, there is currently no consensus in the literature regarding the optimal analgesic regimen after ESS.

   Interestingly, in patients with aspirin-exacerbated respiratory disease (AERD) a triad of asthma, CRS, and aspirin (ASA/NSAID sensitivity), NSAIDs are classically associated with worsening of CRS symptoms. However, cyclooxygenase-2 (COX-2) inhibitors, a selective type of NSAID, have recently been studied as post-ESS analgesics and suggested as possible alternatives to opioids, which have many known potential adverse effects. These agents have also been studied for their anti-inflammatory properties in patients undergoing ESS and have been shown to decrease the levels of circulating prostaglandins in this population. Thus, AERD patients are a particularly important population in which to assess the effect of COX-2 inhibitors on post-operative pain and inflammation. This randomized, prospective study will evaluate both the anti-inflammatory and analgesic effects of a COX-2 inhibitor, celecoxib, in patients with AERD and CRS following endoscopic sinus surgery. The investigators hypothesize that supplementation with celecoxib can potentially improve surgical outcomes and reduce the postoperative usage of opioid analgesics without an increased risk of bleeding or asthma exacerbation.
2. The objectives of this study are: 1) to determine whether the addition of celecoxib to the FESS post-operative analgesia regimen can alter subjective and objective recovery from CRS signs and symptoms, and 2) to determine whether the addition of the COX-2 inhibitor, celecoxib, to the endoscopic sinus surgery post-operative analgesia regimen can reduce the amount of opioid narcotic used by patients for breakthrough pain.
3. Trial Design: The study is a prospective, double-blinded, randomized controlled study and will be conducted at St. Joseph's Hospital in London, ON (CAN). There will be two study arms with 1:1 allocation, one arm will receive the study treatment and the other will receive a placebo;
4. Sample Size Calculation: The initial pre-study sample size was calculated with 80% power at a significance level of 0.05. For the primary objective, previous studies have established that a 40% difference on the Lund-Kennedy Endoscopic Score would be clinically relevant. The statistical power was assumed to be 80%, and the needed significance level (2-tailed alpha error) was assumed to be 5%. Based on the literature, a mean difference of 3.4 and an SD of 2.6 for the Lund-Kennedy endoscopic reporting system was used for calculation, giving a sample size of 22. For the secondary objective, the sample size was calculated as follows. Assuming a difference of 2 of mean pain score (with a standard deviation of 2) on the Numeric Rating scale as significant, a sample size of 16 in each group is required. It has been reported elsewhere a total of 4.5 (+/-4.4) milligram morphine equivalent for patients undergoing a sinus surgery. To reduce this requirement to zero a sample size of 12 in each group would be required. As such, the aim is to enrol 44 patients to account for potential loss of follow-up and ensure the study is appropriately powered.
5. Interventions: Patients in the treatment arm of the study will receive celecoxib 200 mg PO BID for 7 days and patients in the control arm will receive placebo PO BID for 7 days. Both medications are to be started on the evening of the day of surgery. Both groups will also be given a prescription for tramadol, an opioid medication, to be used as needed for breakthrough pain. Specifically, tramadol 50 mg PO Q6H PRN x 10 tablets will be prescribed. Patients will also be permitted to take acetaminophen for breakthrough pain as needed and will be encouraged to use acetaminophen prior to narcotic usage. Finally, all patients will be prescribed a nasal saline rinse which is to be started on postoperative day one.
6. Randomization: Randomization will be via sequential random number generation from 1 to 40. Medications will be prepared by the hospital pharmacy and will be randomized in their preparation by the pharmacy. A master list will be kept in a sealed envelope by the PI in order to break blinding if an emergency occurs. Both study team members and patients will remain blinded to the group until after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older;
* Diagnosis of CRS with nasal polyposis in the setting of AERD, and requiring FESS for management after failing medical management per the Canadian clinical practice guidelines for acute and chronic sinusitis;
* Capable, in the opinion of the primary investigator, of providing informed consent to participate in the study. Participants are required to sign an informed consent form indicating they understand the purpose and nature of the study, and that they are willing to participate.

Exclusion Criteria:

* Known allergies/sensitivities to acetaminophen, opioid, or COX-2 inhibitor NSAIDs
* Inability to read and understand English
* Inability to keep record of exact use of analgesics post-FESS
* History of opioid/narcotic abuse
* Known Ischemic Heart Disease
* Known Mild to moderate congestive heart failure
* Stomach ulceration or bleeding
* Known Inflammatory bowel disease
* Chronic pain or chronic opioid use
* Known renal or hepatic impairment
* Known coagulopathy
* Women who are pregnant or breastfeeding
* Known inability to complete follow-up visits
* Current participation in another clinical trial at time of initial visit
* Use of other medications that impact the serotonin pathway
* Use of medications with potential interactions with celecoxib:

  1. Anticoagulants (warfarin, clopidogrel, dabigatran, enoxaparin)
  2. ACE inhibitors (e.g. captopril, lisinopril)
  3. Diuretics (e.g. furosemide)
  4. Lithium
  5. Cidofovir
  6. Carbamazepine
  7. Antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Post FESS changes in the Lund-Kennedy Endoscopic Score (LKES) | 1 week and 4 weeks post-operatively.
  The postoperative recovery from FESS will be assessed via the changes in the Lund-Kennedy Endoscopic Score (LKES), measured on two time points throughout the post operative recovery.
Post FESS changes in the Peri-Operative Sinus Endoscopy (POSE) score | 1 week and 4 weeks post-operatively.
  The postoperative recovery from FESS will be assessed via the changes in the Peri-Operative Sinus Endoscopy (POSE) score, measured on two time points throughout the post operative recovery.
Post FESS changes in the validated Sino-Nasal Outcome Test 22 (SNOT-22) questionnaire | 1 week and 4 weeks post-operatively.
  The postoperative recovery from FESS will be assessed via the changes in the validated Sino-Nasal Outcome Test 22 (SNOT-22) questionnaire, measured on two time points throughout the post operative recovery.

SECONDARY OUTCOMES:
Post FESS changes in the pain level assessed via the 10-point visual analogue scale | 6h after surgery; 24 hours after surgery; 7 days post-surgery (daily); at the 14th day; and at the 21st day.
  Daily assessment of postoperative pain level via the 10-point visual analogue scale, 6h after surgery, 24h after surgery, daily until day 7, and then at postoperative days 14 and 21.

OTHER OUTCOMES:
Amount of analgesic medication taken on postoperative days 0-7, self reported by the patients. | 0- 7 days post-surgery
  Amount of tramadol, acetaminophen, and any other analgesics taken on postoperative days 0-7, based on patient's self-report.
Number of epistaxis events, self reported by the patients. | 0 to 4 weeks post-surgery
  Assessment of the number of epistaxis events, if they occur, based on patient's self-report, assessed through a 4-week post-op questionnaire.
Compliance with prescribed nasal saline rinses, self reported by the patients. | 0 to 4 weeks post-surgery
  Assessment of the compliance with prescribed nasal saline rinses, based on patient's self-report, assessed through a 4-week post-op questionnaire.
Number of missed days of work/school | 0 to 4 weeks post-surgery
  Assessment of the number of missed days of work/school, based on patient's self-report, assessed through a 4-week post-op questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Sowerby, MD, Principal Investigator — Western University, Canada
Locations (2):
- St. Joseph's Healthcare London, London, Ontario, Canada
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharyya N. Incremental health care utilization and expenditures for chronic rhinosinusitis in the United States. Ann Otol Rhinol Laryngol. 2011 Jul;120(7):423-7. doi: 10.1177/000348941112000701. PMID 21859049
- [Background] Chen Y, Dales R, Lin M. The epidemiology of chronic rhinosinusitis in Canadians. Laryngoscope. 2003 Jul;113(7):1199-205. doi: 10.1097/00005537-200307000-00016. PMID 12838019
- [Background] Blackwell DL, Lucas JW, Clarke TC. Summary health statistics for U.S. adults: national health interview survey, 2012. Vital Health Stat 10. 2014 Feb;(260):1-161. PMID 24819891
- [Background] Xu Y, Quan H, Faris P, Garies S, Liu M, Bird C, Kukec E, Dean S, Rudmik L. Prevalence and Incidence of Diagnosed Chronic Rhinosinusitis in Alberta, Canada. JAMA Otolaryngol Head Neck Surg. 2016 Nov 1;142(11):1063-1069. doi: 10.1001/jamaoto.2016.2227. PMID 27606773
- [Background] Rudmik L, Smith TL, Schlosser RJ, Hwang PH, Mace JC, Soler ZM. Productivity costs in patients with refractory chronic rhinosinusitis. Laryngoscope. 2014 Sep;124(9):2007-12. doi: 10.1002/lary.24630. Epub 2014 Mar 11. PMID 24619604
- [Background] Church CA, Stewart C 4th, O-Lee TJ, Wallace D. Rofecoxib versus hydrocodone/acetaminophen for postoperative analgesia in functional endoscopic sinus surgery. Laryngoscope. 2006 Apr;116(4):602-6. doi: 10.1097/01.MLG.0000208341.30628.16. PMID 16585866
- [Background] Zhao H, Feng Y, Wang Y, Yang B, Xing Z. Comparison of different loading dose of celecoxib on postoperative anti-inflammation and analgesia in patients undergoing endoscopic nasal surgery-200 mg is equivalent to 400 mg. Pain Med. 2011 Aug;12(8):1267-75. doi: 10.1111/j.1526-4637.2011.01196.x. Epub 2011 Aug 3. PMID 21812904
- [Background] Desrosiers M, Evans GA, Keith PK, Wright ED, Kaplan A, Bouchard J, Ciavarella A, Doyle PW, Javer AR, Leith ES, Mukherji A, Schellenberg RR, Small P, Witterick IJ. Canadian clinical practice guidelines for acute and chronic rhinosinusitis. Executive summary. J Otolaryngol Head Neck Surg. 2011 May;40 Suppl 2:S91-8. No abstract available. PMID 21658336
- [Background] Wright ED, Agrawal S. Impact of perioperative systemic steroids on surgical outcomes in patients with chronic rhinosinusitis with polyposis: evaluation with the novel Perioperative Sinus Endoscopy (POSE) scoring system. Laryngoscope. 2007 Nov;117(11 Pt 2 Suppl 115):1-28. doi: 10.1097/MLG.0b013e31814842f8. PMID 18075447